CLINICAL TRIAL: NCT04815096
Title: Imaging Immune Activation in COVID-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CellSight Technologies, Inc. (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20-32477
Record Dates: First submitted 2021-03-23; First posted 2021-03-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: PET-CT Imaging; [18F]F-AraG
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: This is a single center exploratory imaging study involving up to two intravenous microdoses of [18F]F-AraG (the second tracer dose is optional) followed by whole-body PET-CT imaging in participants 18 years of age and older with recent SARS-CoV-2 diagnosis and COVID-19 at least 14 days following onset of symptoms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]F-AraG (Experimental): Radiofluorinated imaging agent, [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine)
  Trade name: VisAcT
  Interventions: Drug: [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine)

INTERVENTIONS:
Drug: [18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D-arabinofuranosylguanine) — [18F]F-AraG is a radiolabeled high affinity substrate for deoxyguanosine kinase (dGK) and a low affinity substrate for deoxycytidine kinase (dCK), which are over-expressed in activated T cells.
  Other Names: VisAcT

SUMMARY:
This is a single center, single arm exploratory imaging study involving up to two intravenous microdoses of [18F]F-AraG (the second tracer dose is optional) followed by whole-body PET-CT imaging in participants with convalescent COVID-19. Up to 80 participants will be enrolled over an accrual period of approximately 48 months.

DETAILED DESCRIPTION:
This is a single center exploratory imaging study involving up to two intravenous microdoses of [18F]F-AraG (the second tracer dose is optional) followed by whole-body PET-CT imaging in participants 18 years of age and older with recent SARS-CoV-2 diagnosis and COVID-19 at least 14 days following onset of symptoms. The primary objective is to determine the anatomical distribution of [18F]F-AraG in participant with convalescent COVID-19 approximately 4 weeks and 1 month to 1 year (optional, 1 month to one year following first PET imaging visit) following onset of symptoms (N = 80). Tracer activity will also be compared with uninfected historical control participants enrolled in prior studies. Up to 80 participants will be enrolled in this study who will be identified in the UCSF LIINC longitudinal COVID-19 cohort study. Each participant will undergo one PET-CT scan following 50 +/- 10 minutes uptake following a single bolus injection of [18F]F-AraG. A second optional [18F]F-AraG dose and PET-CT will be offered approximately 1 month to one year following the initial imaging time point.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Ability to read and understand written informed consent document
* Have a recent diagnosis of SARS-CoV-2 infection as defined by a prior positive SARS-CoV-2 nucleic acid-based diagnostic test performed in a clinical laboratory on one or more nasopharyngeal or respiratory secretion samples.
* > 14 days since onset of COVID-19 symptoms (or if no symptoms, from time of initial nucleic acid based diagnostic test).
* Laboratory evaluations obtained within 60 days prior to entry.

  * Platelet count ≥75,000/mm3
  * ANC >1000/mm3
  * Aspartate aminotransferase (AST) <3 x ULN
  * Alanine aminotransferase (ALT) <3 x ULN
  * Calculated creatinine clearance (CrCl) ≥60 mL/min as estimated by the Cockcroft-
  * Gault equation

Exclusion Criteria:

* Any medical condition that would compromise the imaging acquisition, in the opinion of the investigator
* Participants who are pregnant (female participants of childbearing age will be tested prior to injection of imaging agent at entry visit/initial visit - positive test will exclude from further participation in the study)
* Participants who are breastfeeding
* Female participants of reproductive potential (defined as women who have not been post-menopausal for at least 24 consecutive months (i.e., who have had menses within the preceding 24 months), or women who have not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy) must have a negative urine or serum pregnancy test with a sensitivity of at least 25 mIU/mL performed within 24 hours prior to PET imaging. Females of reproductive potential will need to be on 2 forms of birth control (excluding withdrawal or timing methods).
* Participants who have had prior allogeneic stem cell or solid organ transplant.
* Screening absolute neutrophil count <1,000 cells/mm3, platelet count <75,000 cells/mm3, hemoglobin < 8 mg/dL, estimated creatinine clearance <60 mL/minute, aspartate aminotransferase >3 x ULN, alanine aminotransferase >3 x ULN.
* Known SARS-CoV-2 shedding within 5 days of PET imaging.
* Previously diagnosed myelodysplasia syndrome or history of lymphoproliferative disease prior to study entry
* Active systemic autoimmune diseases not related to COVID-19.
* COVID-19 vaccine prior to the first PET imaging session. Participants may receive COVID-19 vaccination after the first PET imaging session and the optional second PET scan, with the scan being performed at least 2 weeks following the most recent vaccine dose.
* Prior PET scan or therapeutic radiation within 1 year of study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Determine the anatomical distribution of [18F]F-AraG in participant with convalescent COVID-19 greater than 4 weeks (N = 80). Tracer activity will be compared with sex and age-matched uninfected historical control participants enrolled in prior studies. | 4 weeks
  To determine regional uptake of [18F]F-AraG in participants with convalescent COVID-19.

SECONDARY OUTCOMES:
[18F]F-AraG uptake in participants with convalescent COVID-19 over time | 5 months
  To determine the anatomical distribution of [18F]F-AraG in participant with convalescent COVID-19 approximately 4 weeks and 5 months (optional) over time.
Determine if [18F]F-AraG PET-CT is able to detect differences in T cell activation between convalescent COVID-19 participants and age-matched uninfected historical control participants. | 1 year
  Determine if [18F]F-AraG PET-CT is able to detect differences in T cell activation between convalescent COVID-19 participants with and without persistent symptoms (PASC).
Determine if [18F]F-AraG uptake correlates with direct blood measures of immune activation and SARS-CoV-2 specific T cell responses. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Henrich, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No